CLINICAL TRIAL: NCT06071117
Title: EFFECTIVENESS OF VIRTUAL REALITY GLASSES VERSUS WHITE NOISE ON DENTAL ANXIETY IN CHILDREN WITH ATTENTION DEFICIT/ HYPERACTIVITY DISORDER(A RANDOMIZED CONTROLLED CLINICAL TRIAL)
Brief Title: EFFECTIVENESS OF VIRTUAL REALITY GLASSES VERSUS WHITE NOISE ON DENTAL ANXIETY IN CHILDREN WITH ATTENTION DEFICIT/ HYPERACTIVITY DISORDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Nahla Aly, clinical instructor at pediatric dentistry department, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0646-03/2023
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Glasses (VR) (Experimental)
  Interventions: Device: Virtual Reality Glasses (VR)
- White noise (Active Comparator)
  Interventions: Other: White noise
- Basic behavior management techniques (Sham Comparator)
  Interventions: Behavioral: Basic behavior management techniques

INTERVENTIONS:
Device: Virtual Reality Glasses (VR) — Children allocated to this group will be distracted using VR glasses during dental treatment which is an individual headset that has earphones incorporated. Age-appropriate cartoons and movies will be shown to the children. The VR glasses will be then introduced to the children. The children will be given time to accommodate with the device before starting the procedure. The VR glasses will be applied during the dental examination and treatment.
  Arms: Virtual Reality Glasses (VR)
Other: White noise — Wireless kids' headphones will be introduced to the children allocated to this group. They will be given some time to accommodate with the headphones. Then, the white noise will be played and children will be asked to concentrate on the music during the procedure.
  White noise stimulus will be set at 70 decibels, within the "normal conversation" volume range and below what is considered harmful to hearing. The white noise of rain sound, managed with an iPhone application called Muse. The decibel level of white noise will be calibrated using a portable digital sound level meter
  Arms: White noise
Behavioral: Basic behavior management techniques — Children allocated to this group will be managed by the basic behavior guidance techniques: (Tell-Show-Do). No adjunctive distraction tool will be used.
  Arms: Basic behavior management techniques

SUMMARY:
The present study aims to assess and compare the effectiveness of distraction technique using virtual reality glasses and white noise with basic behavior guidance techniques on dental anxiety in children with Attention Deficit/ Hyperactivity Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with ADHD according to the DSM-V criteria and diagnosis confirmed by a pediatric neurologist.
* All children should be on stimulant medication.
* No previous dental experience.
* Written consent of the legal guardian.

Exclusion Criteria:

* Children with physical disabilities or other psychiatric disorders.
* Children with visual or hearing disabilities.
* Patients requiring emergency treatment

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Dental anxiety assessment | up to one week
  This will be assessed using Facial Image Scale (FIS). The FIS comprises one item with a response set of five faces (ranging from a very sad to a very smiley face). Children will be asked to indicate which of the faces they feel most like at that moment, it is a 'state' measure of anxiety that provides an immediate reflection of how the child is feeling.
Pulse rate | up to one week
  The pulse rate will be measured using a pulse oximeter. Normal range is considered from 70-110.
Level of cooperation | up to one week
  Venham's Behavior rating scale (VBRS) will be used to evaluate the overall child's behavior. The changes will be recorded to assess the change in the child's cooperation during the procedure. Venham's Behavior rating scale classifies the child's behavior into 6 categories with scores ranging from 0 to 5. A score of 0 means total cooperation and a score of 5 refers to complete absence of compliance and cooperation and the requirement of physical restraint. The operator will assign a score to each child based on the child's behavior by analysis of the recorded videotape.

CONTACTS AND LOCATIONS:
Overall Officials: Nahla A Aly, BDS, Principal Investigator — Alexandria University; Amina M AbdElrahman, PhD, Study Director — Alexandria University; Karin ML Dowidar, PhD, Study Chair — Alexandria University; Tarek Omar, PhD, Study Director — University of Alexandria
Locations (1):
- Pediatric Neurology Outpatient Clinic, Faculty of Medicine, Alexandria University, Egypt, Alexandria, Egypt